CLINICAL TRIAL: NCT07345793
Title: Mmediate and Short-Term Effects of Dry Needling, Percutaneous Neuromodulation, and Percutaneous Electrolysis on Muscle Tone and Pain: A Two-Phase Randomized Experimental Study in Healthy Subjects and Patients With Chronic Neck Pain.
Brief Title: Effects of Minimally Invasive Techniques in Healthy and Chronic Cervical Pain Individuals
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Carlos Romero Morales, Physiotherapist, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25/787-EC_X
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Chronic Neck Pain
MeSH Terms: interventions — Dry Needling; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This study is designed as a two-phase randomized experimental trial with parallel group assignment.
  In the first phase, healthy volunteers will be randomly assigned to one of three intervention groups:
  1. Dry Needling (DN) - mechanical stimulation of an active myofascial trigger point in the upper trapezius.
  2. Percutaneous Neuromodulation (PENS) - low-frequency electrical stimulation applied near the accessory nerve through an acupuncture needle.
  3. Percutaneous Electrolysis (EPE) - galvanic current (1 mA, three impacts of 5 seconds) applied through a needle at the trigger point.
  All participants will undergo a single treatment session. Assessments of pain intensity (VAS) and muscle mechanical properties (tone, stiffness, elasticity measured by MyotonPRO) will be performed before the intervention, immediately after, and 24 hours later.
  In the second phase, the same study design, intervention parameters, and outcome measures will be applied to a population of patients with chroni
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dry needling (Experimental)
  Interventions: Procedure: Dry needling
- Percutaneous electrical nerve stimulation (Experimental)
  Interventions: Procedure: Percutaneous nerve stimulation
- Percutaneous electrolysis (Experimental)
  Interventions: Procedure: Percutaneous electrolysis

INTERVENTIONS:
Procedure: Dry needling — Dry needling will be performed on the upper trapezius muscle at an active myofascial trigger point. A sterile, single-use solid filament needle (0.30 × 40 mm) will be inserted until eliciting three local twitch responses (LTRs). The needle will then be withdrawn immediately after obtaining the final response. The technique aims to normalize motor endplate activity and reduce local and referred pain through mechanical and neurophysiological modulation.
  Arms: Dry needling
Procedure: Percutaneous nerve stimulation — Percutaneous neuromodulation will be applied using a sterile acupuncture needle (0.30 × 40 mm) inserted near the accessory nerve pathway in the upper trapezius region. A low-frequency alternating current (10 Hz, 250 μs pulse width) will be delivered for 15 minutes using an electrotherapy device approved for clinical use. The objective is to modulate neuromuscular excitability and decrease pain perception through peripheral and central mechanisms.
  Arms: Percutaneous electrical nerve stimulation
Procedure: Percutaneous electrolysis — Percutaneous electrolysis will be performed by inserting a sterile acupuncture needle (0.30 × 40 mm) into the active myofascial trigger point of the upper trapezius. A galvanic current of 1 mA will be applied for three impacts of 5 seconds each using an approved electrolysis device. This technique produces a controlled local inflammatory response, promoting tissue regeneration and analgesia through electrochemical and neurophysiological effects.
  Arms: Percutaneous electrolysis

SUMMARY:
Brief Summary:

This project consists of two sequential experimental phases designed to analyze the immediate and 24-hour effects of three invasive physiotherapy techniques -dry needling (DN), percutaneous neuromodulation (PENS), and percutaneous electrolysis (EPE)- on muscle tone and pain perception.

In the first phase, the study will be conducted on healthy volunteers to assess the physiological responses and safety profile of the interventions under controlled conditions. Each participant will receive one of the three randomly assigned interventions (DN, PENS, or EPE), applied to the upper trapezius muscle. Pain perception (Visual Analog Scale, VAS) and muscle mechanical properties (tone, stiffness, and elasticity) will be measured before and after the intervention, and after 24 hours, using the MyotonPRO device.

In the second phase, the same protocol and parameters will be applied to patients with chronic neck pain, in order to compare the magnitude and persistence of the effects between healthy subjects and symptomatic individuals.

This study aims to improve understanding of the short-term physiological mechanisms of invasive physiotherapy techniques and their relative effectiveness in managing chronic neck pain. The findings will contribute to the development of more precise and evidence-based treatment protocols for musculoskeletal pain.

ELIGIBILITY:
INCLUSION CRITERIA Phase 1 - healthy subjects

1. Age between 18 and 65 years.
2. Healthy individuals without any current musculoskeletal or neurological pathology.
3. Presence of a palpable myofascial trigger point in the upper trapezius muscle.
4. No neck or shoulder pain requiring medical treatment in the past three months.
5. Willingness to refrain from other physiotherapy or manual therapy interventions during the study period.
6. Ability to understand and provide written informed consent

Phase 2 - Patients with Chronic Neck Pain

1. Age between 18 and 65 years.
2. Diagnosis of chronic mechanical or tension-type neck pain lasting for at least 3 months.
3. Presence of at least one active myofascial trigger point in the upper trapezius muscle.
4. Pain intensity between 3 and 7 on a 10-cm Visual Analog Scale (VAS) at baseline.
5. No previous invasive physiotherapy treatments (dry needling, electrolysis, or neuromodulation) within the last 4 weeks.
6. Ability and willingness to attend all study sessions and follow-up assessments.
7. Signed informed consent before participation.

EXCLUSION CRITERIA

1. History of cervical or shoulder surgery.
2. Neurological, systemic, or rheumatologic disorders affecting the cervical or upper limb region.
3. Anticoagulant therapy or known bleeding disorders.
4. Pregnancy or suspected pregnancy.
5. Skin infection, wound, or dermatological condition at or near the intervention site.
6. Use of analgesic, anti-inflammatory, or muscle relaxant medications within 48 hours prior to the intervention.
7. Prior invasive physiotherapy (dry needling, PENS, or EPE) in the target area during the past month.
8. Contraindications to electrical stimulation (for PENS or EPE groups), such as implanted pacemaker or metal implants near the treatment area.
9. Fear of needles (trypanophobia) or intolerance to invasive procedures.
10. Participation in another clinical trial within the past 3 months.
11. Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2026-02-06 (Estimated); Study Completion 2026-02-08 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline (pre-intervention), immediately post-intervention, and 24 hours post-intervention.
  Pain perception will be measured using a 10 cm Visual Analog Scale (VAS), where 0 indicates no pain and 10 indicates worst imaginable pain. Participants will mark their perceived pain intensity at rest. The scale is a reliable and validated tool for assessing subjective pain in musculoskeletal disorders.

SECONDARY OUTCOMES:
Muscle tone | Baseline and immediately post-intervention, and 24 hours post-intervention
  Muscle tone will be assessed using the MyotonPRO device, which measures the natural oscillation frequency (Hz) of the muscle at rest. The upper trapezius will be evaluated at a standardized point corresponding to the active myofascial trigger point region. Higher frequency values indicate increased muscle tone.
Muslce stiffness | Baseline, immediately post intervention and 24 hours post-intervention
  Muscle stiffness will be evaluated using the MyotonPRO, which calculates the muscle's resistance to deformation expressed in newtons per meter (N/m). This parameter reflects the biomechanical rigidity of the tissue.
Muscle elasticity | Baseline, immedialely post intervention and 24 hours post intervention
  Elasticity will be measured with the MyotonPRO, expressed as the logarithmic decrement of the muscle's oscillation. Lower values indicate greater elasticity and better recovery capacity after deformation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fernández-de-Las-Peñas C., Dommerholt J. Myofascial Trigger Points: Pathophysiology and Evidence-Informed Diagnosis and Management. Pain Medicine. 2018.
- [Result] Abat F. et al. Effectiveness of percutaneous electrolysis for tendinopathies. Br J Sports Med. 2015.
- [Result] Rodríguez-Sanz J. et al. Dry Needling in the Management of Musculoskeletal Pain. Brazilian Journal of Physical Therapy. 2014.
- [Result] Pirri C, Manocchio N, Sorbino A, Pirri N, Foti C. Percutaneous Electrolysis for Musculoskeletal Disorders Management in Rehabilitation Settings: A Systematic Review. Healthcare (Basel). 2025 Jul 23;13(15):1793. doi: 10.3390/healthcare13151793. PMID 40805826
- [Result] Hoy D, March L, Woolf A, Blyth F, Brooks P, Smith E, Vos T, Barendregt J, Blore J, Murray C, Burstein R, Buchbinder R. The global burden of neck pain: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1309-15. doi: 10.1136/annrheumdis-2013-204431. Epub 2014 Jan 30. PMID 24482302
- [Result] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284